CLINICAL TRIAL: NCT03113955
Title: A Single-arm Trial of Transcatheter Arterial Chemoembolization With Tandem Microspheres in the Treatment of Localized Hepatocellular Carcinoma
Brief Title: STOPPER CHINA:With Tandem Microspheres in the Treatment of Localized Hepatocellular Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Varian Medical Systems (Industry)
Responsible Party: Sponsor
Organization: Varian, a Siemens Healthineers Company (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2382
Record Dates: First submitted 2017-03-06; First posted 2017-04-14 (Actual); Results first posted 2021-04-19 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Localized Hepatocellular Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single -arm (Experimental): A Single-arm Trial of Transcatheter Arterial Chemoembolization with Tandem Microspheres in the Treatment of Localized Hepatocellular Carcinoma
  Interventions: Device: Tandem Microsphere loaded with Epirubicin

INTERVENTIONS:
Device: Tandem Microsphere loaded with Epirubicin — The primary objective of this study is to evaluate the safety and efficacy of transcatheter arterial chemoembolization with Tandem Microspheres loaded with Epirubicin in the treatment of patients with localized hepatocellular carcinoma (HCC)

SUMMARY:
A Single-arm Trial of Transcatheter Arterial Chemoembolization with Tandem Microspheres in the Treatment of Localized Hepatocellular Carcinoma

DETAILED DESCRIPTION:
It is a prospective, single-arm, multicenter study. The primary effectiveness endpoint for this clinical trial is 6-month overall objective tumor response (ORR).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is able to provide informed consent and must sign the Institutional Review Board/Ethics Committee (IRB/EC) approved Informed Consent Form.
2. Male or female of age ≥18 and ≤75 years.
3. Confirmed diagnosis of HCC according to the diagnostic criteria included in the management guideline issued by China's Ministry of Health in 2017.
4. HCC is diagnosed for the first time or recurrence of tumor after surgical or ablation treatment.
5. Single tumor less than 7cm in diameter or multiple tumors with maximum 3 lesions with >1cm in diameter, individual diameter <7cm and less than 10cm in total diameter.
6. no previous chemotherapy, radiotherapy or transarterial embolization (with or without chemotherapy) for HCC
7. Preserved liver function (Child-Pugh A or B7).
8. ECOG Performance Status 0 or 1.

Exclusion Criteria:

1. Presence of vascular invasion or extra-hepatic spread of disease, or diffuse HCC, defined as >50% liver involvement , or arteriovenuous fistula
2. Macrovascular invasion of main or primary branches of portal vein at entry into the study
3. Any contraindication for TACE treatment
4. Any contraindication for Epirubicin administration
5. Advanced liver disease (bilirubin levels >2 mg/dl, AST or ALT >5 times upper limit of normal)
6. Renal failure or insufficient renal function (Creatinine levels >2 mg/dl)
7. Subject unable to receive MRI examination
8. Pregnant or breast feeding woman, or plan to become pregnant during treatment or within 12 months of treatment
9. couldn't commit reliable birth control measures during treatment or within 12 months of treatment
10. Subject is participating other investigational drug or device clinical trial within 30 days of signing the informed consent
11. Subject is not suitable to participate in the study as judged by investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Peng, Study Director — BSC China
Locations (10):
- China (10):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Guangdong Nanfang Hospital, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Zhongda Hospital Affiliated Southeast University, Nanjing, Jiangsu
  - Shengjing Hospital Affiliated China Medical University, Shenyang, Liaoning
  - Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Second Aff. Hosp. of Zhejiang University College of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang W, Zhang S, Zhong B, Cai W, Gao L, Li B, Yao D, Zhao Y, Sun Z, Zhou S, Zhang T, Chen X, Ju S, Wang YC. Dynamic changes of radiological and radiomics patterns based on MRI in viable hepatocellular carcinoma after transarterial chemoembolization. Abdom Radiol (NY). 2025 May;50(5):2110-2120. doi: 10.1007/s00261-024-04676-z. Epub 2024 Nov 15. PMID 39542948
- [Derived] Zhu HD, Li X, Sun JH, Zhu X, Liu ZY, Li HL, Lu J, Yan ZP, Shao GL, He XF, Chao M, Lu LG, Zhong BY, Li R, Zhang Q, Teng GJ. Transarterial Chemoembolization with Epirubicin-Loaded Microspheres for Hepatocellular Carcinoma: A Prospective, Single-Arm, Multicenter, Phase 2 Study (STOPPER Trial). Cardiovasc Intervent Radiol. 2024 Mar;47(3):325-336. doi: 10.1007/s00270-024-03666-4. Epub 2024 Feb 27. PMID 38413420

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single -Arm
Started | 109
Completed | 92
Not Completed | 17

BASELINE CHARACTERISTICS:
Arm/Group | Single -Arm
Number analyzed (Participants) | 109
Age, Categorical [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: A total of 109 subjects were enrolled, among them one subject coded as 3733S010 was confirmed as cholangiocarcinoma after being enrolled and receiving initial treatment. The subject continuously received follow-up but was not included in the per protocol group for analysis.
  Participants
    number analyzed (Participants) | 108
    <=18 years | 0
    Between 18 and 65 years | 66
    >=65 years | 42
Age, Continuous [Geometric Mean (Standard Deviation); unit: years] — Population: A total of 109 subjects were enrolled, among them one subject coded as 3733S010 was confirmed as cholangiocarcinoma after being enrolled and receiving initial treatment. The subject continuously received follow-up but was not included in the per protocol group for analysis.
  years
    number analyzed (Participants) | 108
    (all) | 60.22 (8.67)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: A total of 109 subjects were enrolled, among them one subject coded as 3733S010 was confirmed as cholangiocarcinoma after being enrolled and receiving initial treatment. The subject continuously received follow-up but was not included in the per protocol group for analysis.
  Participants
    number analyzed (Participants) | 108
    Female | 21
    Male | 87
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: A total of 109 subjects were enrolled, among them one subject coded as 3733S010 was confirmed as cholangiocarcinoma after being enrolled and receiving initial treatment. The subject continuously received follow-up but was not included in the per protocol group for analysis
  Participants
    Han of Chinese: number analyzed (Participants) | 108
    Han of Chinese | 108
Region of Enrollment [Number; unit: participants] — Population: Measure Analysis Population Description: A total of 109 subjects were enrolled, among them one subject coded as 3733S010 was confirmed as cholangiocarcinoma after being enrolled and receiving initial treatment. The subject continuously received follow-up but was not included in the per protocol group for analysis.
  participants
    China: number analyzed (Participants) | 108
    China | 108
Child-Pugh Score [Count of Participants; unit: Participants] — Child-Pugh, classification standard is a commonly used clinically to quantitative assessment of the liver reserve function classification standard. when the Child will be five patient's indicators (including the general situation, ascites, the concentration of serum bilirubin, serum albumin, and prothrombin time) of the different states are divided into three levels, 1 point, 2 and 3 points. Five indicators score together, combined the lowest is 5 points, the highest is 15 points, Class A=5 points, Class B=7-9, Class C=10-15, the higher score, the worse the liver reserve function. Population: A total of 109 subjects were enrolled, among them one subject coded as 3733S010 was confirmed as cholangiocarcinoma after being enrolled and receiving initial treatment. The subject continuously received follow-up but was not included in the per protocol group for analysis.
  Participants
    number analyzed (Participants) | 108
    Class A | 97
    Class B | 11
Disease History [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: A total of 109 subjects were enrolled, among them one subject coded as 3733S010 was confirmed as cholangiocarcinoma after being enrolled and receiving initial treatment. The subject continuously received follow-up but was not included in the per protocol group for analysis.
  Participants
    Diabetes: number analyzed (Participants) | 108
    Diabetes | 16
    Hypertension | 25
    Cirrhosis | 74
    Hepatitis B | 90
    Hepatitis C | 8
ECOG Performance Status [Count of Participants; unit: Participants] — ECOG Performance:
  0 point is fully active, able to carry on all pre-disease performance without restriction; 1 point is restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; 2 points is ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours; 3 points is Capable of only limited self-care, confined to bed or chair more than 50% of waking hours. 4 points is completely disabled. Cannot carry on any self-care. Totally confined to bed or chair. 5 points is dead. Population: Measure Analysis Population Description: A total of 109 subjects were enrolled, among them one subject coded as 3733S010 was confirmed as cholangiocarcinoma after being enrolled and receiving initial treatment. The subject continuously received follow-up but was not included in the per protocol group for analysis.
  Participants
    0 Score: number analyzed (Participants) | 108
    0 Score | 97
    1 Score | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Tumor Response at 6 Months by MRI (Magnetic Resonance Imaging)
Description: The objective response rate measured by MRI used EASL (European Society for the Study of the Liver) and mRECIST (Improved criteria for evaluating the efficacy of solid tumors) , Overall Response (OR) = CR + PR.
  1. Per Response Evaluation Criteria In Solid Tumors Criteria (mRECIST ) for target lesions : Complete Response (CR), Disappearance of any intratumoral arterial enhancement in all target lesions; Partial Response (PR), At least a 30% decrease in the sum of the diameters of viable (enhancement in the arterial phase) target lesions, taking as reference the baseline sum of the diameters of target lesions.
  2. Per Response Evaluation Criteria In Solid Tumors Criteria (EASL) for target lesions: Complete Response (CR), Disappearance of all known disease and no new lesions determined by two observations not less than 4 weeks apart; Partial Response (PR), At least 50% reduction in total tumor load of all measurable lesions determined by two observations not less than 4 weeks apart.
Time Frame: At 6 months
Population: Total enrolled 109 subjects , 7 subjects were not completed 6 months primary endpoint follow up visit and were not included in the per protocol group for analysis. So overall Number of Participants Analyzed were 102.
Measure: Number; unit: participants
Arm/Group | Single -Arm
Number analyzed (Participants) | 102
participants
  6-month ORR (EASL criteria) | 75
  6-month ORR (mRECIST criteria) | 73

2. Secondary Outcome: Kaplan-Meier Analyses the Percent of Participants for Time to Progression (TTP) at 12 Months
Description: Kaplan-Meier analyses the percent of participants for TTP which is defined as the length of time from the treatment initiation to either the date of the first disease progression occurred, as assessed by the investigators, or the date of the subject died due to any cause, whichever comes earlier. EASL and mRECIST response assessment of target lesion for HCC. TTP (also referred as "time to treatment failure") will be measured by a few data items list below:
  * The date of the disease progression in the Overall Response form
  * The date of lost-to-follow due to:
    * Adverse events
    * Progressive disease/insufficient therapeutic response
    * Death
    * Failure to return
    * Refusing treatment/being unwilling to cooperate/withdrawing consent
  * The very last date by scanning all available dates in the database
  * The desired cut-off days
Time Frame: At 12 months
Population: Measure Analysis Population Description: Measure Analysis Population Description: A total of 109 subjects were enrolled, among them one subject coded as 3733S010 was confirmed as cholangiocarcinoma after being enrolled and receiving initial treatment. The subject continuously received follow-up but was not included in the per protocol group for analysis.
Measure: Number; unit: Percent of participants
Arm/Group | Single -Arm
Number analyzed (Participants) | 108
Percent of participants
  EASL: number analyzed (Participants) | 73
  EASL | 10
  mRECIST: number analyzed (Participants) | 72
  mRECIST | 8

3. Secondary Outcome: Number of Participants With Objective Tumor Response at 30-day
Description: as for outcome 1
Time Frame: At 1month
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Single -Arm
Number analyzed (Participants) | 108
Participants
  EASL Response | 86
  mRECIST Response | 86

4. Secondary Outcome: Kaplan-Meier Analyses the Percent of Participants for PPF(Proportion Progression-Free) at 12 Months
Description: Kaplan-Meier analyses the percent of participants for PPF which is defined as the length of time from the treatment initiation, that treated subjects are still progression-free. EASL and mRECIST response assessment of target lesion for HCC.
  The data items to be captured will include:
  * The date of the disease progression in the Overall Response form
  * The very last date by scanning all available dates in the database
  * The desired cut-off days The proportion of any time point will be determined by the Kaplan-Meier estimates.
Time Frame: from first TACE to 12 months
Population: as for outcome 2
Measure: Number; unit: Percent of participants
Arm/Group | Single -Arm
Number analyzed (Participants) | 108
Percent of participants
  EASL: number analyzed (Participants) | 73
  EASL | 10
  mRECIST: number analyzed (Participants) | 72
  mRECIST | 8

5. Secondary Outcome: Kaplan-Meier Analyses the Percent of Participants for Overall Survival
Description: Kaplan-Meier analyses the percent of participants for Overall survival which is defined as the length of time from the treatment initiation, that treated subjects are still alive. The Kaplan-Meier analysis is aimed to capture the all-cause death for each subject. Subjects who are lost-to-follow will be considered being censored.
  There are three critical data items to be captured:
  * Death date
  * The very last date in the database (e.g. follow-up visit date and/or site reported AE date)
  * The desired cut-off days (e.g. 6-month OS at 182 days, 12-month OS at 365 days) In addition to the Kaplan-Meier survival curve, the median survival time (mOS) will also be used to represent the study cohort.
Time Frame: from first TACE to 12 months
Population: Measure Analysis Population Description: Measure Analysis Population Description: A total of 109 subjects were enrolled, among them one subject coded as 3733S010 was confirmed as cholangiocarcinoma after being enrolled and receiving initial treatment, 1 subject withdrew consent from study participation at 6 month, 1 subject withdrew consent from study participation at 12 month. All 3 subjects are not included in the group for overall survival analysis.
Measure: Number; unit: Percent of participants
Arm/Group | Single -Arm
Number analyzed (Participants) | 106
Percent of participants | 100

6. Secondary Outcome: Number of Adverse Events Relate to Study Device in 12 Months Post Procedure
Description: Number and documents of adverse events relate to study device in 12 months post procedure
Time Frame: in 12 months
Population: as for outcome 2
Measure: Number; unit: adverse events
Arm/Group | Single -Arm
Number analyzed (Participants) | 108
adverse events
  SAEs of related with TANDEM Microspheres | 17
  Non-serious AEs of related with TANDEM Microspheresrate | 301

7. Secondary Outcome: Number of Participants With Objective Tumor Response at 3 Months
Description: as for outcome 1
Time Frame: At 3 months
Population: Total enrolled 109 subjects , 4 subjects were not completed 3 months primary endpoint follow up visit and were not included in the per protocol group for analysis. So overall Number of Participants Analyzed were 105.
Measure: Count of Participants; unit: Participants
Arm/Group | Single -Arm
Number analyzed (Participants) | 105
Participants
  EASL Response | 84
  mRECIST Response | 85

8. Secondary Outcome: Kaplan-Meier Analyses the Percent of Participants for Time to Extrahepatic Spread
Description: Kaplan-Meier analyses the percent of participants for Time to Extrahepatic Spread which the length of time from the treatment initiation to the development of extrahepatic spread of the disease via imaging assessment.
  The data items to be considered will include:
  * The date of the extrahepatic spread in the Overall Response form
  * The very last date by scanning all available dates in the database
  * The desired cut-off days
Time Frame: At 12 month
Population: as for outcome 2
Measure: Number; unit: Percent of participants
Arm/Group | Single -Arm
Number analyzed (Participants) | 108
Percent of participants | 20

ADVERSE EVENTS:
Time Frame: 12 months
Description: Measure Analysis Population Description: Measure Analysis Population Description: A total of 109 subjects were enrolled, among them one subject coded as 3733S010 was confirmed as cholangiocarcinoma after being enrolled and receiving initial treatment. The subject continuously received follow-up but was not included in the per protocol group for analysis.
Arm/Group | Single -Arm
All-Cause Mortality (participants affected / at risk) | 7/108
Serious Adverse Events (participants affected / at risk) | 13/108
Other Adverse Events (participants affected / at risk) | 75/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single -Arm (N=108)
Liver abscess (Hepatobiliary disorders) | 5 (6) — There was 6 cases of hepatic abscess reported in the per protocol group
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hepatic cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Jaundice hepatocellular (Hepatobiliary disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Post embolisation syndrome (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single -Arm (N=108)
Investigations (Blood and lymphatic system disorders) | 23 (81)
Gastrointestinal disorders (Gastrointestinal disorders) | 27 (48)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 60 (91)
General disorders and administration site conditions (General disorders) | 14 (18)
Hepatobiliary disorders (Hepatobiliary disorders) | 14 (20)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 6 (6)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 7 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-03-23): https://cdn.clinicaltrials.gov/large-docs/55/NCT03113955/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-28): https://cdn.clinicaltrials.gov/large-docs/55/NCT03113955/SAP_001.pdf